CLINICAL TRIAL: NCT02500043
Title: Randomized, Double-blind, Phase 3 Study Evaluating TAS-102 Plus Best Supportive Care (BSC) Versus Placebo Plus BSC in Patients With Metastatic Gastric Cancer Refractory to Standard Treatments
Brief Title: Study of TAS-102 or Placebo Plus BSC in Patients With Metastatic Gastric Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TO-TAS-102-302; 2015-002683-16 (EudraCT Number)
Record Dates: First submitted 2015-07-13; First posted 2015-07-16 (Estimated); Results first posted 2021-09-16 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Refractory Metastatic Gastric Cancer
Keywords: Gastric Cancer; Metastatic Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — trifluridine tipiracil drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TAS-102+BSC (Experimental): Participants received 35 milligrams per meter square (mg/m^2) of TAS-102 tablets orally twice daily (BID) for 5 days per week (i.e., from Days 1 to 5 and Days 8 to 12) for 2 weeks followed by 14 days rest in each 28-day cycle along with BSC until a discontinuation criterion (participant withdrawal, disease progression, irreversible treatment-related Grade 4 non-hematologic event, physician's decision, pregnancy or death) was met.
  Interventions: Drug: TAS-102
- Placebo+BSC (Experimental): Participants received 35 mg/m^2 of matching placebo for TAS-102 tablets orally BID for 5 days per week (i.e., from Days 1 to 5 and Days 8 to 12) for 2 weeks followed by 14 days rest in each 28-day cycle along with BSC until discontinuation criterion (participant withdrawal, disease progression, irreversible treatment-related Grade 4 non-hematologic event, physician's decision, pregnancy or death) was met.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAS-102 — 35 mg/m2/dose of TAS-102 orally, twice daily on days 1-5 and days 8-12 of each 28-day cycle.
  Arms: TAS-102+BSC
Drug: Placebo — 35 mg/m2/dose of placebo orally, twice daily on days 1-5 and days 8-12 of each 28-day cycle.
  Arms: Placebo+BSC

SUMMARY:
The purpose of this trial is to compare the effects of TAS-102 and best supportive care (BSC) with Placebo (an inactive drug) and best supportive care on metastatic gastric cancer.

DETAILED DESCRIPTION:
This is a multinational, double-blind, two-arm, parallel, randomized, Phase 3 study evaluating the efficacy and safety of TAS-102 plus BSC versus placebo plus BSC in participants with metastatic gastric cancer who have previously received at least 2 prior regimens for advanced disease. Eligible participants will be centrally randomized (2:1) to TAS-102 + BSC (experimental arm) or placebo + BSC (control arm).

ELIGIBILITY:
Inclusion Criteria:

1. Has histologically confirmed non-resectable, metastatic gastric adenocarcinoma including adenocarcinoma of the gastroesophageal junction.
2. Has previously received at least 2 prior regimens for advanced disease and were refractory to or unable to tolerate their last prior therapy.
3. Has measureable or nonmeasurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.
4. Is able to take medications orally (ie, no feeding tube).
5. Has an Eastern Cooperative Oncology Group performance status of 0 or 1.
6. Has adequate organ function as defined by protocol defined labs.
7. Women of childbearing potential must have a negative pregnancy test and must agree to adequate birth control if conception is possible. Males must agree to adequate birth control.

Exclusion Criteria:

1. Has certain serious illnesses or medical conditions
2. Has had certain other recent treatment e.g. major surgery, anticancer therapy, extended field radiation, received investigational agent within the specified time frames prior to study drug administration.
3. Has previously received TAS-102.
4. Has unresolved toxicity of greater than or equal to Common Terminology Criteria for Adverse Events Grade 2 attributed to any prior therapies.
5. Is a pregnant or lactating female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 507 (Actual)
Dates: Start 2016-02-24 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2019-12-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (139):
- United States (24):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - St. Jude Heritage Healthcare, Fullerton, California
  - Los Angeles Cancer Network, Los Angeles, California
  - University of Southern California - Keck School of Medicine, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - 21st Century Oncology, Jacksonville, Florida
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Illinois CancerCare P.C., Peoria, Illinois
  - University of Kentucky, Lexington, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - Dartmouth-Hitchcock Medical Center (DHMC), Lebanon, New Hampshire
  - Laura & Isaac Perlmutter Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Univeristy of Rochester Medical Center, Rochester, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Pittsburgh Medical Cancer Center, Pittsburgh, Pennsylvania
  - Roger Williams Medical Center, Providence, Rhode Island
  - Coastal Bend Cancer Center, Corpus Christi, Texas
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Belarus (3):
  - Gomel Regional Clinical Oncology Dispensary, Homyel
  - Minsk City Clinical Oncology Dispensary, Minsk
  - Republican center for oncology and medical radiology n.a. Alexandrov, Minsk
- Belgium (4):
  - Clinique universitaire Saint Luc, Brussels
  - Grand Hopital de Charleroi, Charleroi
  - University Hospital Antwerpen, Edegem
  - UZ Leuven, Leuven
- Recherche GCP Research, Montreal, Canada
- Czechia (5):
  - Fakultni Nemocniceu sv. Anny v Brne, Brno
  - Faculty Hospital Hradec Kralove, Hradec Králové
  - Fakultní Nemocnice Olomouc, Olomouc
  - Nemocnice Na Homolce, Prague
  - VFN Praha, Prague
- France (11):
  - ICO Paul Papin, Angers
  - Centre Léon Bérard, Lyon
  - Hopital de La Timone, Marseille
  - Hôpital Saint Joseph, Marseille
  - Centre Val D'Aurelle, Montpellier
  - Hopital Europeen Georges Pompidou, Paris
  - AP-HP - HU La Pitié-Salpêtrière - Charles-Foix, Paris
  - Hôpital Saint-Jean, Perpignan
  - Centre medico-chirurgical Magellan, Pessac
  - Centre Eugène Marquis, Rennes
  - Centre René Gauducheau, Saint-Herblain
- Germany (7):
  - Technische Universitaet Muenchen, Munich, Bavaria
  - Charite Universitaetsmedizin Berlin, Berlin
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Staedtisches Krankenhaus Muenchen Neuperlach, München
  - Leopoldina-Krankenhaus, Schweinfurt
  - Universitaetsklinikum Ulm, Ulm
- Ireland (3):
  - St James Hospital, Dublin
  - The Adelaide and Meath Hospital, Dublin, Incorporating The National Children's Hospital, Dublin
  - Waterford Regional Hospital, Waterford
- Israel (7):
  - Soroka Medical Centre, Beersheba
  - Rambam healthcare campus, Haifa
  - Wolfson Medical Center, Holon
  - Hadassah Ein Karem, Jerusalem
  - Rabin MC Belinson Hospital, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Ramat Gan
- Italy (15):
  - IRCCS Centro di Riferimento Oncologico - Aviano, Aviano (PN)
  - Humanitas Gavazzeni, Bergamo
  - Fondazione Poliambulanza Istituto Ospedaliero, Brescia
  - Struttura Complessa di Oncologia, Cremona
  - Azienda Ospedaliero - Universitaria Careggi, Florence
  - Azienda Ospedaliera San Martino, Genova
  - IRCCS - Istituto Scientifico Romagnolo Per lo Studio e la Cura Dei Tumori (I.R.S.T.), Meldola (FC)
  - Istituto Europeo di Oncologia (IEO), Milan
  - A.O. Ospedale 'Niguarda Ca Granda', Milan
  - A.O.U. Seconda Universita'degli Studi di Napoli, Napoli
  - A.O.U. San Luigi Gonzaga, Orbassano (TO)
  - Azienda Ospedaliero Universitaria Pisana (AOUP), Pisa
  - A.O.R. San Carlo, Potenza
  - Istituto Clinico Humanitas, Rozzano (Mi)
  - A.O. della Valtellina e della Valchiavenna Ospedale di Sondrio, Sondrio
- Japan (9):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Gunma Prefectural Cancer Center, Ōta, Gunma
  - Ibaraki Prefectural Central Hospital, Kasama, Ibaraki
  - Osaka National Hospital, Osaka, Osaka
  - Osaka General Medical Center, Osaka, Osaka
  - Sakai City Medical Center, Sakai, Osaka
  - Tochigi Cancer Center, Utsunomiya, Tochigi
  - Toyama University Hospital, Tōyama, Toyama
  - Iwate Medical University, Morioka
- Poland (6):
  - Górnoslaskie Centrum Medyczne im. prof. Leszka Gieca, Katowice
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Regionalny Osrodek Onkologiczny, Lodz
  - Szpital MSWiA i Warminsko - Mazurskim Centrum Onkologii w Olsztynie, Olsztyn
  - Opolskie centrum Onkologii, Opole
  - Maria Sklodowska-Curie Memorial Cancer Center, Institute of Oncology, Warsaw
- Portugal (9):
  - Unidade Local de Saúde de Matosinhos E.P.E.- H. Pedro Hispano, Matosinhos Municipality, Porto District
  - Hospital Garcia de Orta, E.P.E., Almada, Setúbal District
  - SNS - Hospital Braga, Braga
  - Fundação Champalimaud, Lisbon
  - Hospital da Luz, S.A., Lisbon
  - Centro Hospitalar do Porto, E.P.E, Porto
  - Instituto Português de Oncologia do Porto Francisco Gentil, E.P.E., Porto
  - Centro Hospitalar de São João, EPE, Porto
  - Centro Hospitalar de Tras-os-Montes e Alto Douro, EPE, Vila Real
- Romania (2):
  - Centrul De Oncologie "Sfantul Nectarie", Craiova, Dolj
  - Spitalul Judetean de Urgenta "Sfantul Ioan cel Nou" Suceava, Suceava
- Russia (7):
  - N.N. Blokhin Russian Cancer Research Center, Moscow
  - Nizhegorodsky Regional Oncology Center, Nizhny Novgorod
  - Budget Institution of Healthcare Omsk Region -Clinical Oncology Dispensary, Omsk
  - North-Western State Medical University n.a. I.I. Mechnikov, Saint Petersburg
  - N.N.Petrov Research Institute of Oncology, Saint Petersburg
  - Saint-Petersburgskiy Oncologic Hospital, Saint Petersburg
  - Republican Oncology Center, Ufa
- Spain (7):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Morales Meseguer, Murcia
  - Hospital Universitario Central de Asturias, Oviedo
  - Corporacio Parc Tauli, Sabadell
- Turkey (Türkiye) (11):
  - Baskent University Adana Practice and Research Centre Kisla, Adana
  - Ankara University Medical Faculty Cebeci Hospital, Ankara
  - Hacettepe University, Ankara
  - Dr. Abdurrahman Yurtaslan Ankara Oncology Training and Research, Ankara
  - Diskapi Yildirim Beyazit Training and Research Hospital, Ankara
  - Uludag University Medical Faculty, Bursa
  - Trakya University Medical Faculty Hospital, Edirne
  - Istanbul Üniversitesi, Istanbul
  - Bezmialem Vakif Üniversitesi Tip Fakültesi Hastanesi, Istanbul
  - Marmara University Pendik Training and Research Hospital, Istanbul
  - Dokuz Eylul University Oncology Institute, Izmir
- United Kingdom (8):
  - East and North Hertfordshire NHS Trust, Northwood, Middlesex
  - NHS Grampian, Aberdeen, Scotland
  - Belfast Health and Social Care Trust - Belfast City Hospital, Belfast
  - Leicester Royal Infirmary, Leicester
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Sarah Cannon Research Institute, London
  - The Christie NHS Foundation Trust, Manchester
  - The Royal Marsden NHS Foundation Trust, Sutton

REFERENCES:
- [Derived] Ying T, Xia R, Zhang Y, Dai J, Wang Y, Xie X. Cost-effectiveness analysis of trifluridine/tipiracil in the treatment of heavily pretreated metastatic gastric cancer from the perspective of Chinese healthcare system. BMJ Open. 2024 Nov 7;14(11):e080846. doi: 10.1136/bmjopen-2023-080846. PMID 39510786
- [Derived] Shitara K, George B, Taieb J, Sundar R, Fakih MG, Makris L, Benhadji KA, Ghidini M. Effects of prior therapies on outcomes with trifluridine/tipiracil in patients with metastatic gastric/gastroesophageal junction cancer in a randomized phase III trial (TAGS). J Cancer Res Clin Oncol. 2023 Sep;149(11):9361-9374. doi: 10.1007/s00432-023-04813-z. Epub 2023 May 22. PMID 37213030
- [Derived] Tabernero J, Alsina M, Shitara K, Doi T, Dvorkin M, Mansoor W, Arkenau HT, Prokharau A, Ghidini M, Faustino C, Gorbunova V, Zhavrid E, Nishikawa K, Ando T, Yalcin S, Van Cutsem E, Sabater J, Skanji D, Leger C, Amellal N, Ilson DH. Health-related quality of life associated with trifluridine/tipiracil in heavily pretreated metastatic gastric cancer: results from TAGS. Gastric Cancer. 2020 Jul;23(4):689-698. doi: 10.1007/s10120-020-01053-9. Epub 2020 Mar 4. PMID 32128634
- [Derived] Ilson DH, Tabernero J, Prokharau A, Arkenau HT, Ghidini M, Fujitani K, Van Cutsem E, Thuss-Patience P, Beretta GD, Mansoor W, Zhavrid E, Alsina M, George B, Catenacci D, McGuigan S, Makris L, Doi T, Shitara K. Efficacy and Safety of Trifluridine/Tipiracil Treatment in Patients With Metastatic Gastric Cancer Who Had Undergone Gastrectomy: Subgroup Analyses of a Randomized Clinical Trial. JAMA Oncol. 2020 Jan 1;6(1):e193531. doi: 10.1001/jamaoncol.2019.3531. Epub 2020 Jan 9. PMID 31600365
- [Derived] Shitara K, Doi T, Dvorkin M, Mansoor W, Arkenau HT, Prokharau A, Alsina M, Ghidini M, Faustino C, Gorbunova V, Zhavrid E, Nishikawa K, Hosokawa A, Yalcin S, Fujitani K, Beretta GD, Cutsem EV, Winkler RE, Makris L, Ilson DH, Tabernero J. Trifluridine/tipiracil versus placebo in patients with heavily pretreated metastatic gastric cancer (TAGS): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2018 Nov;19(11):1437-1448. doi: 10.1016/S1470-2045(18)30739-3. Epub 2018 Oct 21. PMID 30355453
- [Derived] Bando H, Doi T, Muro K, Yasui H, Nishina T, Yamaguchi K, Takahashi S, Nomura S, Kuno H, Shitara K, Sato A, Ohtsu A. A multicenter phase II study of TAS-102 monotherapy in patients with pre-treated advanced gastric cancer (EPOC1201). Eur J Cancer. 2016 Jul;62:46-53. doi: 10.1016/j.ejca.2016.04.009. Epub 2016 May 19. PMID 27208903

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at study centers in 17 countries. Participants were involved in the study from 24 February 2016 to 19 December 2019.
Pre-assignment Details: Overall, 625 participants were screened, of which 118 were screen failures due to inclusion/exclusion criteria not met and 507 were randomized and treated with TAS-102 or placebo along with Best supportive care (BSC) (BSC was given to prevent, control, or relieve complications and side effects with the intention to maximize quality of life (QoL) without a specific antineoplastic regimen).
Period: Overall Study
Arm/Group | TAS-102+BSC | Placebo+BSC
Started | 337 | 170
As-Treated (AT) Population (All participants who received at least 1 dose of study treatment.) | 335 | 168
Completed | 0 | 0
Not Completed | 337 | 170
Not completed — Randomized, but not Treated | 2 | 2
Not completed — Ongoing at Date of Cut-Off | 19 | 3
Not completed — Adverse Event | 33 | 11
Not completed — Clinical Progression | 54 | 35
Not completed — Radiological Progression | 192 | 110
Not completed — Physician's Decision | 11 | 3
Not completed — Withdrawal by Subject | 14 | 4
Not completed — Death | 11 | 2
Not completed — Protocol Deviation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on the Intent-to-Treat (ITT) population that included all randomized participants, regardless of whether or not study treatment was administered.
Groups:
- TAS-102+BSC: Participants received 35 mg/m^2 of TAS-102 tablets orally BID for 5 days per week (i.e., from Days 1 to 5 and Days 8 to 12) for 2 weeks followed by 14 days rest in each 28-day cycle along with BSC until a discontinuation criterion (participant withdrawal, disease progression, irreversible treatment-related Grade 4 non-hematologic event, physician's decision, pregnancy or death) was met.
- Total: Total of all reporting groups
Arm/Group | TAS-102+BSC | Placebo+BSC | Total
Number analyzed (Participants) | 337 | 170 | 507
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.8 (10.78) | 62.0 (10.04) | 62.5 (10.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 53 | 138
  Male | 252 | 117 | 369
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 244 | 113 | 357
  Black/African American | 1 | 2 | 3
  Asian | 51 | 29 | 80
  Not collectable | 38 | 24 | 62
  Other | 3 | 2 | 5
European Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — The ECOG performance status was used to evaluate participant's disease progression and the effect of the disease on the participant's activities of daily living. It ranged on the scale from 0-5 (0 equal to [=] normal activity; 1= symptoms but ambulatory; 2= in bed for less than (<) 50 percent (%) of the time; 3= in bed for greater than (>) 50% of the time; 4= 100% bedridden; 5= dead). Time to definitive deterioration in ECOG performance status score from baseline was defined as change from 0, 1 to greater than or equal to (>=2), or from 2 to >=3.
  Participants
    ECOG Grade 0 | 123 | 68 | 191
    ECOG Grade 1 | 214 | 102 | 316

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death due to any cause. Participants without documented death were censored at last follow-up or cut-off date, whichever comes first. OS was estimated by Kaplan-Meier method.
Time Frame: From the date of randomization to the data cut-off date (maximum duration: up to approximately 46 months)
Population: Analysis was performed on the ITT population that included all randomized participants, regardless of whether or not study treatment was administered.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TAS-102+BSC | Placebo+BSC
Number analyzed (Participants) | 337 | 170
months | 5.7 [4.8 to 6.2] | 3.6 [3.1 to 4.1]
Statistical Analysis 1: Comparison: TAS-102+BSC vs Placebo+BSC; TAS-102+BSC and Placebo+BSC were compared using the stratified log-rank test using the 3 randomization stratification factors (region, ECOG performance status, and prior treatment with ramucirumab). The hazard ratio was estimated using a stratified Cox's proportional hazard (CPH) model and survival was summarized using Kaplan Meier estimates; Test type: Other; p = 0.0003, Log Rank — One-sided P-Value; Hazard Ratio (HR) = 0.6917, 95% CI 2-sided [0.5597 to 0.8548]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from randomization until the date of first occurrence of investigator-assessed radiological disease progression or death due to any cause, whichever came first. Disease progression as per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) for target lesions were defined as target lesions with at least 20 % relative increase in the sum of diameters with reference to the smallest sum on study, including the baseline sum and this sum demonstrated an absolute increase of at least 5 millimeter (mm) or the appearance of one or more new lesions or Unequivocal progression of existing non-target lesions. All alive participants with no disease progression as of the analysis cut-off date were censored at the last tumor assessment. PFS was estimated by Kaplan-Meier method.
Time Frame: From the date of randomization to the cut-off date (maximum duration: up to approximately 46 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TAS-102+BSC | Placebo+BSC
Number analyzed (Participants) | 337 | 170
months | 2.0 [1.9 to 2.3] | 1.8 [1.7 to 1.9]
Statistical Analysis 1: Comparison: TAS-102+BSC vs Placebo+BSC; TAS-102+BSC and Placebo+BSC were compared using the stratified log-rank test using the 3 randomization stratification factors (region, ECOG performance status, and prior treatment with ramucirumab). The hazard ratio was estimated using a stratified CPH model and survival was summarized using Kaplan Meier estimates; Test type: Other; Hazard Ratio (HR) = 0.5723, 95% CI 2-sided [0.4674 to 0.7008]

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAE)
Description: Any untoward medical condition that occurs in a participants while participating in a clinical study and does not necessarily have a causal relationship with the use of the study medication was considered an adverse event (AE). A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. TEAEs/TESAEs were defined as events that started on or after treatment or started before treatment and worsened after the start of treatment through 30 days after the last dose of study treatment.
Time Frame: From the first dose of study treatment until 30 days after the last dose of study treatment (maximum duration: up to approximately 46 months)
Population: Analysis was performed on the As-treated (AT) population that included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | TAS-102+BSC | Placebo+BSC
Number analyzed (Participants) | 335 | 168
Participants
  TEAE | 319 | 151
  TESAE | 143 | 70

4. Other Pre Specified Outcome: Overall Response Rate (ORR)
Description: Overall response rate was defined as the percentage of participants with objective evidence of complete response (CR) or partial response (PR).
  CR was defined as the disappearance of all target or non-target lesions. Any pathological lymph nodes for target lesions or all lymph nodes for non-target lesions were non-pathological morphologically that was reduced in size in short axis to < 10 mm.
  PR was defined as target lesions with at least 30% decrease in the sum of diameters, taking baseline sum diameters as reference.
Time Frame: From the date of randomization to the cut-off date (maximum duration: up to approximately 46 months), assessed every 8 weeks
Population: Analysis was performed on tumor response (TR) population that included participants in the ITT population that met 2 criteria: had measurable disease (at least 1 target lesion) at baseline; had at least 1 post-baseline evaluation or early disease progression/cancer-related death occurred before first evaluation on treatment (post-baseline).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAS-102+BSC | Placebo+BSC
Number analyzed (Participants) | 290 | 145
percentage of participants | 4.5 [2.4 to 7.5] | 2.1 [0.4 to 5.9]

5. Other Pre Specified Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the proportion of participants with a best overall response of complete response (CR), partial response (PR), or stable disease (SD). The assessment of DCR was based on Investigator review of radiologic images and following RECIST criteria (version 1.1, 2009).
Time Frame: as for outcome 4
Population: Analysis was performed on TR population that included participants in the ITT population that met 2 criteria: had measurable disease (at least 1 target lesion) at baseline; had at least 1 post-baseline evaluation or early disease progression/cancer-related death occurred before first evaluation on treatment (post-baseline).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAS-102+BSC | Placebo+BSC
Number analyzed (Participants) | 290 | 145
percentage of participants | 44.1 [38.3 to 50.1] | 14.5 [9.2 to 21.3]

6. Other Pre Specified Outcome: Time to Deterioration of European Cooperative Oncology Group (ECOG) Performance Status Score From Baseline
Description: The ECOG performance status was used to evaluate participant's disease progression and the effect of the disease on the participant's activities of daily living. It ranges on the scale from 0-5 (0 = normal activity; 1= symptoms but ambulatory; 2= in bed for < 50% of the time; 3= in bed for > 50% of the time; 4= 100% bedridden; 5= dead). Time to definitive deterioration in ECOG performance status score from baseline was defined as a change from 0, 1 to >=2, or from 2 to >=3.
Time Frame: At the time of randomization (Day 1 Cycle 1) and within 24 hours prior to start of study treatment in every cycle (maximum duration: up to approximately 46 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TAS-102+BSC | Placebo+BSC
Number analyzed (Participants) | 337 | 170
months | 4.3 [3.7 to 4.7] | 2.3 [2.0 to 2.8]

7. Other Pre Specified Outcome: Change From Baseline in Quality of Life European Organization for Research and Treatment for Cancer (EORTC) QoL Questionnaire Core 30 (QLQ-C30 Score): Global Health Status
Description: EORTC-QLQ-C30 is a cancer-specific instrument with 30 questions for evaluation of new chemotherapy and provides an assessment of participant reported outcome dimensions. First 28 questions used 4-point scale (1=not at all,2=a little,3=quite a bit,4=very much) for evaluating 5 functional scales (physical,role,emotional,cognitive,social), 3 symptom scales (fatigue,nausea/vomiting,pain) and other single items. For each item,high score represented high level of symptomatology/problem. Last 2 questions represented participant's assessment of overall health and QoL, coded on 7-point scale (1=very poor to 7=excellent). EORTC QLQ-C30 observed values and change from baseline for global health status (scoring of questions 29 and 30) and 5 functional scales, 3 symptom scales and other single items (scoring of questions 1 to 28). Answers were converted into grading scale, with values between 0 and 100. A high score represented a favorable outcome with a best QoL for participant.
Time Frame: Baseline, Day 1 Cycle 2 up to end of treatment (EOT) (within 30 days of last study treatment) and 30-Day safety follow-up visit (maximum duration: up to approximately 46 months)
Population: Analysis was performed on the ITT population that included all randomized participants, regardless of whether or not study treatment was administered. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TAS-102+BSC | Placebo+BSC
Number analyzed (Participants) | 337 | 170
units on a scale
  Cycle 1: number analyzed (Participants) | 279 | 127
  Cycle 1 | -2.7 (17.56) | -5.9 (22.20)
  Cycle 2: number analyzed (Participants) | 187 | 58
  Cycle 2 | -5.9 (20.51) | -7.3 (25.80)
  Cycle 3: number analyzed (Participants) | 121 | 23
  Cycle 3 | -4.1 (18.26) | -1.4 (22.00)
  Cycle 4: number analyzed (Participants) | 79 | 15
  Cycle 4 | -3.6 (17.54) | -1.7 (22.32)
  Cycle 5: number analyzed (Participants) | 55 | 9
  Cycle 5 | -5.9 (18.05) | 11.1 (18.16)
  Cycle 6: number analyzed (Participants) | 36 | 8
  Cycle 6 | -8.8 (23.05) | 15.6 (21.10)
  Cycle 7: number analyzed (Participants) | 28 | 5
  Cycle 7 | -9.5 (21.96) | 20.0 (4.56)
  Cycle 8: number analyzed (Participants) | 23 | 5
  Cycle 8 | -4.3 (23.82) | 16.7 (11.79)
  Cycle 9: number analyzed (Participants) | 14 | 3
  Cycle 9 | 2.4 (17.12) | 16.7 (16.67)
  Cycle 10: number analyzed (Participants) | 11 | 2
  Cycle 10 | -14.4 (25.57) | 25.0 (11.79)
  Cycle 11: number analyzed (Participants) | 5 | 2
  Cycle 11 | -16.7 (37.27) | 25.0 (11.79)
  Cycle 12: number analyzed (Participants) | 2 | 1
  Cycle 12 | -8.3 (11.79) | 33.3
  Cycle 13: number analyzed (Participants) | 1 | 1
  Cycle 13 | 0.0 | 33.3
  Cycle 14: number analyzed (Participants) | 0 | 1
  Cycle 14 |  | 33.3
  Cycle 15: number analyzed (Participants) | 0 | 1
  Cycle 15 |  | 33.3
  Last Collection Cycle: number analyzed (Participants) | 283 | 128
  Last Collection Cycle | -8.8 (20.91) | -9.8 (25.34)
  Safety Follow-Up: number analyzed (Participants) | 39 | 14
  Safety Follow-Up | -16.5 (23.45) | -8.9 (18.33)

8. Other Pre Specified Outcome: EORTC Quality of Life Questionnaire - Gastric-specific Module (EORTC QLQ-STO22): Percentage of Participants With Overall Compliance
Description: The Quality of Life Questionnaire Stomach Cancer Module 22 (QLQ-STO22) assessed symptoms and treatment-related side effects commonly reported in participants. There are 22 questions which comprise 5 scales (dysphagia, dietary restrictions, pain QS22, reflux, and anxiety) and 4 single items (dry mouth, hair loss, taste problems, body image). Most questions use 4-point scale (1='Not at all', 2=a little, 3=quite a bit and 4='Very much'). A linear transformation was used to standardize all scores and single-items to a scale of 0 to 100, where higher score=better level of functioning or greater degree of symptoms.
Time Frame: Baseline, Cycle 1 Day 1 up to end of treatment (EOT) (within 30 days of last study treatment) (maximum duration: up to approximately 46 months)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | TAS-102+BSC | Placebo+BSC
Number analyzed (Participants) | 337 | 170
percentage of participants
  Dysphagia | 86.6 | 78.2
  Dietary Restrictions | 86.6 | 78.2
  Pain QS22 | 86.6 | 78.2
  Reflux | 86.6 | 78.2
  Anxiety | 86.6 | 78.2
  Dry Mouth | 86.4 | 78.2
  Body Image | 85.8 | 78.2
  Hair Loss | 86.6 | 78.2
  Taste Problems | 86.6 | 78.2

ADVERSE EVENTS:
Time Frame: From first dose of study treatment up to 30 days of last study treatment (maximum duration: up to approximately 46 months).
Description: Analysis was performed on the AT population.
Arm/Group | TAS-102+BSC | Placebo+BSC
All-Cause Mortality (participants affected / at risk) | 252/335 | 141/168
Serious Adverse Events (participants affected / at risk) | 143/335 | 70/168
Other Adverse Events (participants affected / at risk) | 319/335 | 151/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAS-102+BSC (N=335) | Placebo+BSC (N=168)
Anaemia (Blood and lymphatic system disorders) | 13 (13) | 4 (5)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 4 (5) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 7 (7) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-Respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 8 (8) | 6 (6)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 3 (4) | 7 (7)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 6 (6) | 2 (2)
Gastric haemorrhage (Gastrointestinal disorders) | 3 (3) | 3 (3)
Gastric stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (6) | 1 (1)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2)
Haematemesis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (3) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 4 (4) | 3 (4)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ulcerative gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 9 (9) | 1 (2)
Asthenia (General disorders) | 1 (1) | 3 (3)
Disease progression (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0)
General physical health deterioration (General disorders) | 21 (25) | 15 (20)
Malaise (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Performance status decreased (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 1 (2) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 0 (0) | 1 (2)
Jaundice (Hepatobiliary disorders) | 2 (2) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Biliary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (2) | 0 (0)
Infection (Infections and infestations) | 2 (3) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 4 (6) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 4 (4) | 2 (2)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 3 (3) | 0 (0)
Typhoid fever (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bilirubin conjugated increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Alkalosis hypochloraemic (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 11 (11) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Ureteric cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 2 (2) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAS-102+BSC (N=335) | Placebo+BSC (N=168)
Anaemia (Blood and lymphatic system disorders) | 142 (249) | 30 (52)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 57 (116) | 3 (14)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 20 (42) | 8 (21)
Neutropenia (Blood and lymphatic system disorders) | 128 (312) | 6 (9)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (3) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 32 (45) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 6 (6) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (3) | 2 (2)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 3 (4) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 13 (15) | 9 (9)
Abdominal pain (Gastrointestinal disorders) | 50 (75) | 27 (34)
Abdominal pain lower (Gastrointestinal disorders) | 3 (3) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 22 (27) | 14 (15)
Anal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal pruritus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 16 (24) | 10 (18)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 44 (53) | 25 (31)
Diarrhoea (Gastrointestinal disorders) | 73 (118) | 24 (28)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 4 (4)
Dyschezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 5 (7) | 3 (4)
Dysphagia (Gastrointestinal disorders) | 14 (16) | 6 (6)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 2 (2)
Flatulence (Gastrointestinal disorders) | 2 (4) | 2 (2)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastric stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (5) | 2 (2)
Haematemesis (Gastrointestinal disorders) | 3 (4) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intra-Abdominal fluid collection (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 3 (3) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 123 (201) | 53 (64)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophageal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 15 (17) | 3 (3)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 80 (104) | 34 (48)
Asthenia (General disorders) | 65 (97) | 37 (45)
Catheter site pain (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 3 (3) | 1 (1)
Chills (General disorders) | 4 (6) | 0 (0)
Drug intolerance (General disorders) | 1 (1) | 0 (0)
Early satiety (General disorders) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 1 (1)
Facial pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 87 (136) | 35 (41)
Feeling abnormal (General disorders) | 1 (1) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 3 (3) | 3 (4)
Hyperthermia (General disorders) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 9 (16) | 8 (8)
Mucosal inflammation (General disorders) | 8 (11) | 3 (3)
Non-Cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 8 (8) | 2 (2)
Oedema peripheral (General disorders) | 17 (17) | 12 (12)
Pain (General disorders) | 5 (6) | 8 (8)
Performance status decreased (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 23 (37) | 8 (9)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 10 (10) | 3 (5)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (2) | 0 (0)
Jaundice (Hepatobiliary disorders) | 2 (2) | 2 (2)
Liver disorder (Hepatobiliary disorders) | 4 (6) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Autoimmune disorder (Immune system disorders) | 0 (0) | 1 (2)
Perfume sensitivity (Immune system disorders) | 1 (1) | 0 (0)
Angular cheilitis (Infections and infestations) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 3 (3) | 0 (0)
Cystitis (Infections and infestations) | 3 (4) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Gingival abscess (Infections and infestations) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1)
Herpes virus infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 3 (4) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (5) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 6 (6) | 2 (2)
Pneumonia (Infections and infestations) | 4 (4) | 1 (1)
Pyuria (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Rhinitis (Infections and infestations) | 3 (3) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 2 (3) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 8 (9) | 0 (0)
Urinary tract infection (Infections and infestations) | 9 (15) | 4 (4)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 3 (4)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Radiation injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase (Investigations) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 16 (17) | 8 (8)
Aspartate aminotransferase (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 21 (26) | 13 (15)
Bilirubin conjugated increased (Investigations) | 1 (2) | 1 (1)
Blood alkaline phosphatase (Investigations) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 30 (35) | 14 (15)
Blood bilirubin (Investigations) | 1 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 17 (27) | 7 (9)
Blood bilirubin unconjugated increased (Investigations) | 1 (2) | 1 (1)
Blood creatinine decreased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 10 (11) | 6 (11)
Blood iron decreased (Investigations) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 7 (9) | 7 (8)
Creatinine renal clearance decreased (Investigations) | 1 (1) | 0 (0)
Enzyme level increased (Investigations) | 2 (2) | 0 (0)
Gamma-Glutamyltransferase increased (Investigations) | 4 (6) | 5 (6)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 2 (2) | 0 (0)
Hepatic enzyme increased (Investigations) | 3 (4) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (7) | 0 (0)
Neutrophil count (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 50 (139) | 1 (1)
Platelet count decreased (Investigations) | 28 (43) | 6 (11)
Platelet count increased (Investigations) | 0 (0) | 1 (1)
Protein total decreased (Investigations) | 2 (2) | 0 (0)
Red blood cell count decreased (Investigations) | 2 (2) | 0 (0)
Red cell distribution width increased (Investigations) | 1 (1) | 0 (0)
Vital capacity abnormal (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 20 (21) | 12 (13)
Weight increased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 23 (59) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 109 (164) | 49 (54)
Dehydration (Metabolism and nutrition disorders) | 4 (6) | 2 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Feeding intolerance (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 9 (10) | 5 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (3) | 3 (5)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 21 (28) | 10 (11)
Hypocalcaemia (Metabolism and nutrition disorders) | 9 (11) | 1 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 9 (11) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 7 (7) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (6) | 7 (8)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 25 (31) | 9 (10)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Bone swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 2 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (2)
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Agnosia (Nervous system disorders) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 8 (10) | 4 (4)
Dysgeusia (Nervous system disorders) | 11 (17) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 6 (8) | 4 (5)
Lethargy (Nervous system disorders) | 2 (2) | 3 (3)
Monoplegia (Nervous system disorders) | 0 (0) | 1 (1)
Myoclonus (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 4 (4) | 1 (1)
Paraesthesia (Nervous system disorders) | 8 (8) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 5 (5) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 2 (2) | 2 (2)
Anxiety (Psychiatric disorders) | 9 (9) | 4 (4)
Confusional state (Psychiatric disorders) | 2 (3) | 3 (3)
Delirium (Psychiatric disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 3 (5) | 2 (2)
Disturbance in social behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Drug abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 11 (12) | 10 (10)
Nervousness (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (4) | 1 (1)
Albuminuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Choluria (Renal and urinary disorders) | 2 (2) | 0 (0)
Dysuria (Renal and urinary disorders) | 5 (5) | 3 (3)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Leukocyturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Microalbuminuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Micturition disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic discomfort (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 6 (7)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 (24) | 16 (16)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 4 (4)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 12 (14) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Palmar-Plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (9) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (4)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Xeroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1)
Embolism (Vascular disorders) | 2 (2) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 7 (7) | 1 (1)
Pallor (Vascular disorders) | 2 (4) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-05-05): https://cdn.clinicaltrials.gov/large-docs/43/NCT02500043/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/43/NCT02500043/SAP_001.pdf